CLINICAL TRIAL: NCT05643378
Title: Role and Outcome of Endovascular Revacularization of Chronic Limb Threatening Ischaemia in Patients With Chronic Kidney Diseases
Brief Title: Role and Outcome of Endovascular Revascularization of Chronic Limb Ischaemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Abdelmohsen Mostafa Osman (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Abdelmohsen Mostafa Osman, principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: endovascular treatment
Record Dates: First submitted 2022-11-26; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Limb Ischemia, Critical
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
identify the safety and efficacy of percutaneous transluminal angioplasty in critical limb ischaemia patients with chronic kidney dieases

DETAILED DESCRIPTION:
patients with chronic kidney diseases are at higher risk of developing peripheral artery diseases needing revascularization of diseased arteries via endovascular transluminal angioplasty

ELIGIBILITY:
Inclusion Criteria:

* all patients with chronic kidney diseases on medical treatment or on dialysis and have critical limb ischaemia

Exclusion Criteria:

* patients with acute renal failure and lower limb ischaemia.
* chronic kidney diseased patients underwent previous intervention or surgery for lower limb ischaemia.
* patients presented with acute limb ischaemia

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients fulfilled these criteria will be included in this study as an availability sample for year duration sample size : 100 patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
one year evaluation for maintaining vessel patency without restenosis or need for re intervention in 100 participants | baseline
  all patients will be scheduled for follow up visits every 3 months for 1 year assessing primary patency and major adverse limb events.
  duplex scanning will be performed for all patients

REFERENCES:
- [Background] Dayama A, Tsilimparis N, Kolakowski S, Matolo NM, Humphries MD. Clinical outcomes of bypass-first versus endovascular-first strategy in patients with chronic limb-threatening ischemia due to infrageniculate arterial disease. J Vasc Surg. 2019 Jan;69(1):156-163.e1. doi: 10.1016/j.jvs.2018.05.244. PMID 30579443
- [Background] Imamura T. Optimal therapeutic strategy for those with chronic kidney disease and peripheral artery disease receiving peripheral vascular intervention. Clin Cardiol. 2020 Dec;43(12):1348. doi: 10.1002/clc.23483. Epub 2020 Oct 19. No abstract available. PMID 33073876
- [Background] Moussa Pacha H, Al-Khadra Y, Darmoch F, Soud M, Mamas MA, Moussa Pacha A, Zaitoun A, Kaki A, AlJaroudi WA, Alraies MC. In-hospital outcome of peripheral vascular intervention in dialysis-dependent end-stage renal disease patients. Catheter Cardiovasc Interv. 2020 Feb 15;95(3):E84-E95. doi: 10.1002/ccd.28522. Epub 2019 Oct 21. PMID 31631511